CLINICAL TRIAL: NCT01823042
Title: A Randomized, Controlled, Open-label Study to Assess the the Efficacy of Enteral Nutrition in Fill of the Treatment Blank Period of the Postoperative Maintain Remission Medication for Crohn's Disease (CD).
Brief Title: The Efficacy of Enteral Nutrition in Fill of the Treatment Blank Period of the Postoperative Maintain Remission Medication for Crohn's Disease (CD)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jinling Hospital, China (Other)
Responsible Party: Principal Investigator, Zhu Weiming, vice director of General surgery institute, Jinling Hospital, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDS-2
Record Dates: First submitted 2013-03-25; First posted 2013-04-04 (Estimated); Last update posted 2013-04-04 (Estimated); Status verified 2013-03

CONDITIONS: Crohn's Disease
Keywords: Crohn's Disease; maintain remission; postoperative recurrence; surgery; living quality
MeSH Terms: conditions — Crohn Disease | interventions — Azathioprine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- enteral nutrition+azathioprine (Experimental): Patients is fasting and receive enteral nutrition and azathioprine treatment.
  Interventions: Drug: azathioprine+enteral nutrition
- azathioprine (Experimental): Patients have regular diet and receive only azathioprine treatment.
  Interventions: Drug: Azathioprine

INTERVENTIONS:
Drug: azathioprine+enteral nutrition
  Arms: enteral nutrition+azathioprine
Drug: Azathioprine
  Arms: azathioprine

SUMMARY:
Crohn's disease(CD) is a agnogenic disease which has a lifelong relapse tendency even after surgery treatment.So maintain remission medications were routinely given to patients after surgery.But maintain remission medications,as azathioprine,6-MP, ciclosporin,tripterygium glycosides, had a onset time.The therapeutic effect may appear 3 months~6months after taken medicine.There is a treatment blank period between surgery and onset time of maintain remission medications.Enteral nutrition has been used in the induction remission and maintain remission for CD.May be it can fill the treatment blank period.

DETAILED DESCRIPTION:
Crohn's disease(CD) is a agnogenic disease which has a lifelong relapse tendency even after surgery treatment.So maintain remission medications were routinely given to patients after surgery.But maintain remission medications,as azathioprine,6-MP, ciclosporin,tripterygium glycosides, had a onset time.The therapeutic effect may appear 3 months~6months after taken medicine.There is a treatment blank period between surgery and onset time of maintain remission medications.Enteral nutrition has been used in the induction remission and maintain remission for CD.May be it can fill the treatment blank period.

ELIGIBILITY:
Inclusion Criteria:

* Subjects should have a definitive diagnosis of Crohn's disease, based on WHO criteria
* Subjects having curative resection/ileocolonic anastomosis，pathologically diagnosed as Crohn's disease
* Lesions located in ileum or ileocecal region
* Males and females ≥ 18 years old, including women who are not pregnant or lactating at the time of enrollment.
* Body weight between 40 and 100 kg, inclusive.
* Subjects should have a CDAI score <150 at week 0
* Able to swallow tablets
* Are capable of providing written informed consent and obtained at the time of enrollment
* Willing to adhere to the study visit schedule and other protocol requirements.

Exclusion Criteria:

* Bacterial,viral or other microbial infection(including HIV)
* any of the following medications taken within 12 weeks before surgery: cyclosporine, tacrolimus, sirolimus, mycophenolate mofetil, or other investigational drugs
* any of ongoing therapy for Crohn's disease with: 5-ASA compounds, steroids, immune modifiers, systemic antibiotics, and tube feeding
* Needing orally administered corticosteroids for the treatment of other diseases. Inhaled or dermatologic preparations are acceptable.
* Previous or current use of infliximab.
* current use of prescription doses or chronic/frequent use of NSAIDs
* Treatment with narcotic pain medications. (Anti-diarrheal agents such as loperamide and diphenoxylate are permitted, providing that the dose is not increased during the study period.)
* History of pancreatitis, except for subjects with a known but removed cause(such as gallstone pancreatitis)
* WBC <3.0 x 109/L, hemoglobin <80 g/L, Platelets<50,000/mm3 at the time of enrollment (or within the previous 6 months, if known)
* History of abnormal liver function tests, including AST or ALT >1.5 times upper limit of normal, alkaline phosphatase >2 times upper limit of normal, total bilirubin >2.5 mg/dL at screening (or within the previous 6 months, if known)
* With short bowel syndrome (defined as requiring oral or parenteral supplemental or total nutrition to maintain stable body weight, or more than 100 cm of small bowel resected)
* History of malignancy
* Women who are pregnant or lactating at the time of enrollment, or who intend to be during the study period.
* Participation in other clinical trial within the past 6 months

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2012-10; Primary Completion 2013-07 (Estimated); Study Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
The change of patients'CDAI. | at 0 week, the 4 weeks, the 8 weeks, the 12weeks
patients' endoscopic score(Rutgeerts score). | at the 12weeks

SECONDARY OUTCOMES:
The change of haematological inflammation marker(CRP,ESR) | at 0 week, the 4 weeks, the 8 weeks, the 12weeks
The change of patients'IBDQ. | at 2 week, the 6 weeks, the 12 weeks
The change of blood routine examination and blood biochemistry. | at 0 week,4 weeks,8 weeks,12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- General Surgery Institute,Jinling Hospital, Nanjing, Jiangsu, China